CLINICAL TRIAL: NCT02950142
Title: The Effect of Evidence-based Order Sets Within a CPOE System on the Quantity and Quality of Laboratory Test Ordering in Family Practice: a Cluster Randomised Trial
Brief Title: Evidence-based Laboratory Test Order Sets in Primary Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: KU Leuven (Other); University Ghent (Other); Norwegian Institute of Public Health (Other Government); Sciensano (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: S59472; CB1611 (Other: Belgian Health Care Knowledge Centre)
Record Dates: First submitted 2016-10-25; First posted 2016-10-31 (Estimated); Last update posted 2020-01-23 (Actual); Status verified 2020-01

CONDITIONS: Diabetes Mellitus; Hypertension; Cardiovascular Diseases; Fatigue; Anemia; Liver Diseases; Medication Monitoring; Gout; Chronic Kidney Diseases; Lung Embolism; Acute Coronary Syndrome; Diarrhea; Thyroid Diseases; Sexually Transmitted Diseases; Rheumatoid Arthritis; Obesity; General Check-up
Keywords: order sets; decision support; laboratory test; primary care
MeSH Terms: conditions — Diabetes Mellitus; Hypertension; Cardiovascular Diseases; Fatigue; Anemia; Liver Diseases; Gout; Renal Insufficiency, Chronic; Pulmonary Embolism; Acute Coronary Syndrome; Diarrhea; Thyroid Diseases; Sexually Transmitted Diseases; Arthritis, Rheumatoid; Obesity | interventions — Medical Order Entry Systems

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CPOE with order sets (Experimental): Physicians who use CPOE including order sets for large range of indications.
  Interventions: Other: CPOE with order sets for lab testing
- CPOE without order sets (Active Comparator): Physicians who use CPOE without order sets.
  Interventions: Other: CPOE without order sets for lab testing

INTERVENTIONS:
Other: CPOE with order sets for lab testing — CPOE including series of recommended tests ordered per indication
  Other Names: CPOE with order sets for laboratory testing
  Arms: CPOE with order sets
Other: CPOE without order sets for lab testing — CPOE only
  Other Names: CPOE without order sets for laboratory testing
  Arms: CPOE without order sets

SUMMARY:
Cluster randomised controlled trial to evaluate what the effect is of evidence-based order sets aimed at five indications on the appropriateness of laboratory test ordering in primary care.

DETAILED DESCRIPTION:
Cluster randomised controlled trial in Belgian primary care practices. Participants will be primary care physicians working in primary care practices affiliated to one of three collaborating laboratories in the Leuven, Ghent or Antwerp regions.

Primary care practices will be allocated and randomized to either the intervention or control group. Physicians in PCPs randomized to the intervention will be offered order sets based on indication when using the CPOE for ordering laboratory tests. The effect of order sets will be analyzed for 17 common indications for ordering laboratory tests in Belgian primary care: diabetes mellitus, hypertension, cardiovascular disease, general check-up, unexplained fatigue, anemia, liver pathology, medication monitoring, gout, chronic kidney disease, lung embolism, acute coronary syndrome, diarrhea, thyroid disease, sexually transmitted disease, rheumatoid arthritis and obesity.

ELIGIBILITY:
Inclusion Criteria:

* Primary care practices will be considered eligible if all the physicians active in the practice agree to be involved in the study
* All family physicians will be considered eligible if they:

  * Collaborate with either MCH, Anacura or AML for their laboratory test orders
  * Agree to use the online CPOE for their laboratory test orders
  * Use a computerized EHR for patient care
  * Agree to the terms in the informed consent

Exclusion Criteria:

* Primary care practices where one or more physicians refuse to be enrolled will be excluded

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 288 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2018-06-01 (Actual); Study Completion 2019-08-01 (Actual)

PRIMARY OUTCOMES:
Appropriateness | 3 months
  number of appropriate tests for 17 study indications

SECONDARY OUTCOMES:
Missed or delayed diagnoses | 1 year
  Incidence of missed or delayed diagnoses after laboratory test
Laboratory test volume | 1 year
  Total volume of ordered laboratory tests

OTHER OUTCOMES:
Downstream or cascade clinical activities | 1 year
  All downstream or cascade clinical activities as a result of abnormal test result

CONTACTS AND LOCATIONS:
Locations (1):
- Academic Centre for General Practice, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: No
IPD sharing plan not yet decided. Decision will be made upon start of trial.

REFERENCES:
- [Background] Delvaux N, De Sutter A, Van de Velde S, Ramaekers D, Fieuws S, Aertgeerts B. Electronic Laboratory Medicine ordering with evidence-based Order sets in primary care (ELMO study): protocol for a cluster randomised trial. Implement Sci. 2017 Dec 6;12(1):147. doi: 10.1186/s13012-017-0685-6. PMID 29212546
- [Derived] Piessens V, Delvaux N, Heytens S, Aertgeerts B, De Sutter A. Downstream activities after laboratory testing in primary care: an exploratory outcome of the ELMO cluster randomised trial (Electronic Laboratory Medicine Ordering with evidence-based order sets in primary care). BMJ Open. 2022 Apr 4;12(4):e059261. doi: 10.1136/bmjopen-2021-059261. PMID 35379642
- [Derived] Delvaux N, Piessens V, Burghgraeve T, Mamouris P, Vaes B, Stichele RV, Cloetens H, Thomas J, Ramaekers D, Sutter A, Aertgeerts B. Clinical decision support improves the appropriateness of laboratory test ordering in primary care without increasing diagnostic error: the ELMO cluster randomized trial. Implement Sci. 2020 Nov 4;15(1):100. doi: 10.1186/s13012-020-01059-y. PMID 33148311

DOCUMENTS (2):
  • Study Protocol: Full protocol (2017-08-07): https://cdn.clinicaltrials.gov/large-docs/42/NCT02950142/Prot_000.pdf
  • Statistical Analysis Plan (2019-07-18): https://cdn.clinicaltrials.gov/large-docs/42/NCT02950142/SAP_001.pdf